CLINICAL TRIAL: NCT00224302
Title: Treatment of Major Depressive Episodes During the Course of Psychotic Disorders With Duloxetine
Brief Title: Treatment of MDEs During the Course of Psychotic Disorders With Duloxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Duloxetine-Zink
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2005-09

CONDITIONS: Psychotic Disorders
Keywords: Schizophrenia,; schizoaffective disorder,; major depressive episode,; combination,; duloxetine
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
We evaluate the efficacy and tolerability of duloxetine in the treatment of major depressive episodes during the course of psychotic disorders

DETAILED DESCRIPTION:
Major depressive episodes (MDE) frequently occur during the course of schizophrenic psychoses, both as as "post-psychotic" depressions, and also independently from psychotic episodes. A number of clinical studies reported the application of different antidepressive substances, such as Imipramine, Reboxetine or Venlafaxine. In general, the treatment of schizophrenic patients with antidepressive drugs can be considered as necessary and save, resulting in therapeutic guidelines of different psychiatric societies. However, since 5 to 10 % of the schizophrenic patients commit suicide, there is still much effort necessary in order to improve the treatment of affective symptoms in schizophrenic psychoses.The recently introduced antidepressive substance Duloxetine selectively inhibits as a SSNRI the reuptake of serotonine and noradrenaline from the synaptic cleft. Duloxetine was proven as antidepressive, anxiolytic and analgetic in a series of multi-centre, placebo-controlled investigations. Based on these considerations and on successful experiences in single case reports we aim to investigate the therapeutic effects of duloxetine in patients with lifetime diagnoses of the schizophrenic spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode, Severity: CDSS at least 8 points or HAMD at least 15 points, indication for the treatment with duloxetine
* Lifetime diagnosis of a psychotic disorder (PANSS positive scale below 15 points)
* Age between 18 and 65,
* Informed consent

Exclusion Criteria:

* No informed consent,
* Contraindications with respect to duloxetine,
* Gravidity or missing anticonceptive safety
* Substance dependance (excluded nicotin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
CDSS, HAMD, PANSS, SANS

SECONDARY OUTCOMES:
PANSS, SANS, Serum levels of antipsychotic substances, Body weight, EPMS,Prolactin, blood pressure, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Zink, MD, Principal Investigator — Central Institute of Mental Health, Department of Psychiatry, Mannheim, Germany
Locations (1):
- Central Institute of Mental Health, Department of Psychiatry,, Mannheim, Baden-Wurttemberg, Germany